CLINICAL TRIAL: NCT01084772
Title: A Multicenter, Randomized, Clinical Outcome of VISIONAIRE™ Patient Matched Technology vs. Standard Surgical Instrumentation in Total Knee Arthroplasty
Brief Title: Visionaire™ Versus Standard Instrumentation Safety and Efficacy in Total Knee Arthroplasty (TKA)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VISSTD01
Record Dates: First submitted 2010-02-19; First posted 2010-03-10 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Degenerative Arthritis of Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VISIONAIRE Instrumentation (Other): TKA with VISIONAIRE instrumentation
  Interventions: Other: VISIONAIRE Total Knee Arthroplasty
- Standard Instrumentation (Other): TKA with standard instrumentation
  Interventions: Other: Standard Total Knee Arthroplasty

INTERVENTIONS:
Other: VISIONAIRE Total Knee Arthroplasty — TKA will be performed with VISIONAIRE instrumentation, depending on randomization assignment.
  Arms: VISIONAIRE Instrumentation
Other: Standard Total Knee Arthroplasty — TKA will be performed with standard instrumentation, depending on randomization assignment.
  Arms: Standard Instrumentation

SUMMARY:
The objective of this study is to assess outcomes following TKA, utilizing two surgical techniques. Patients will be randomized to one of two arms: TKA with standard instrumentation and TKA with VISIONAIRE™ patient-matched cutting blocks. Data will be collected at preoperative, operative/discharge, 3 months, 1 year and 2 years after TKA. The secondary objective of this study is to compare the safety, quality of life, and economic outcomes of TKA when these two techniques are utilized. This study does not involve treatment or investigational products, as all components are FDA cleared and are commercially available.

DETAILED DESCRIPTION:
This is a prospective study comparing VISIONAIRE™ to standard TKA instrumentation. The objective of this study is to evaluate the safety and efficacy of TKA using VISIONAIRE™ when compared with standard instrumentation, including device survival, improvement in function and implant alignment after TKA. This study will also document any device-related, surgical complications and/or adverse radiographic observations.

In contrast with the control group clinical outcomes following TKA completed with VISIONAIRE™ have yet to be assessed. The current investigation will determine if there is any difference in TKA outcomes when VISIONAIRE™ patient matched technology is utilized versus standard instrumentation. All patients meeting the inclusion/exclusion criteria specified in this protocol will be asked to participate in the study. If the patient consents to participate, they will be enrolled in the study and randomized to one of the two study arms. Patients requiring TKA will be implanted with Legion, Genesis II or Journey BCS (Smith & Nephew) total knee implant systems. Standard instrumentation will be used to assist the surgeon in placing the implant in the control group. In the VISIONAIRE™ group, standard instrumentation will not be used in the surgery. Patients randomized to the VISIONAIRE™ arm will have an MRI preoperatively that will be used to create the customized cutting blocks. All patients will have an x-ray at each postoperative interval.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the inclusion criteria.

1. Patient diagnosed with degenerative arthritis of the knee requiring a unilateral primary TKA.
2. Patient is of legal age to consent and is skeletally mature.
3. Patient is willing to sign and date an ethics-approved consent form.
4. Patient is willing to be available for two-year follow-up postoperatively

Exclusion Criteria:

Patients must not meet any of the exclusion criteria.

1. Patient is known to have poor bone stock making a TKA unjustifiable.
2. Patient is immuno-suppressed.
3. Patient has physical, emotional or neurological conditions that would compromise the patient's compliance with postoperative rehabilitation and follow-up.
4. Patient is pregnant or may become pregnant during the course of the study.
5. Patient has a history of prior ipsilateral major knee surgery (e.g. arthroplasty, high tibial osteotomy, or tibial plateau fracture). Minor prior procedures such as ACL repair, meniscectomy, or arthroscopy are not excluded.
6. Patient has active, localized or systemic infection.
7. Patient is severely overweight (BMI >40).
8. Patient is a prisoner.
9. Subject has a significant MRI (magnetic resonance imaging) exclusion or contraindication.
10. Patient has had a total joint arthroplasty of the contralateral limb in the last 12 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2012-06-21 (Actual); Primary Completion 2014-04-15 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beate Hanson, MD, PhD, Study Director — Smith & Nephew, Inc.
Locations (7):
- United States (6):
  - Orthopaedic Surgery Specialist, Ltd., Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Town & Country Orthopedics, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Slocum Research & Education Foundation, Eugene, Oregon
- Malabar Orthopaedic Clinic, Windsor, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to enroll 196 subjects; 134 subjects were recruited to the study prior to its termination due to insufficient total enrollment. Subjects were enrolled from 21 June 2012 to 15 April 2014. Early termination was approved May 2014 and sites were officially notified of study termination in September 2015.
Groups:
- VISIONAIRE Instrumentation: TKA with VISIONAIRE instrumentation
  Total Knee Arthroplasty: TKA was performed with VISIONAIRE instrumentation. Total knee arthroplasty was performed using customized surgical instruments created from preoperative imaging and specialized software, VISIONAIRE Patient-Matched Technology, which was used to match the patient's unique anatomy.
- Standard Instrumentation: TKA with standard instrumentation
  Total Knee Arthroplasty was performed using conventional instrumentation.
Period: Baseline
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Started | 68 | 66
Completed | 61 | 60
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 7 | 6
Period: 3 Months
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Started | 61 | 60
Completed | 58 | 58
Not Completed | 3 | 2
Not completed — Death | 1 | 0
Not completed — Study Termination | 2 | 2
Period: 1 Year
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Started | 58 | 58
Completed | 55 | 50
Not Completed | 3 | 8
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Study Termination | 0 | 7
Period: 2 Years
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Started | 55 | 50
Completed | 46 | 46
Not Completed | 9 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 5 | 2
Not completed — Study Termination | 3 | 2

BASELINE CHARACTERISTICS:
Population: There were 134 participants; however, demographic data for 1 participant was marked "lost" in the database.
Groups:
- Total: Total of all reporting groups
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation | Total
Number analyzed (Participants) | 68 | 65 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (8.71) | 67.5 (7.70) | 68.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 77
  Male | 28 | 28 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Not Hispanic | 52 | 46 | 98
  Black, Not Hispanic | 2 | 3 | 5
  Hispanic | 1 | 0 | 1
  Other | 0 | 1 | 1
  Aus-Asian | 1 | 1 | 2
  Aus-Caucasian | 12 | 14 | 26
Height [Mean (Standard Deviation); unit: cm] | 168.0 (9.84) | 168.0 (10.12) | 168.0 (9.94)
Weight [Mean (Standard Deviation); unit: kg] | 88.3 (17.80) | 83.7 (17.77) | 86.1 (17.86)

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Clinical (KSS) Score at 2 Years Following Surgery - Total Score
Description: The KSS was used to rate both the prosthesis function and the patient's functional abilities after TKA. The KSS Total Score (0-100 points) included a combined evaluation of joint motion (0-25 points), instability (0-25 points), alignment (0-25 points), and symptoms (0-25 points). A higher score indicated a better outcome for subjects.
Time Frame: 2 years postoperatively
Population: The Knee Society Clinical Score was not completed for all enrolled subjects. Data was only available for 83 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 42 | 41
score on a scale | 91.4 (13.7) | 94.3 (8.9)

2. Primary Outcome: Knee Society Clinical (KSS) Score at 2 Years Following Surgery - Clinical Evaluation Questionnaire
Description: The KSS was used to rate both the prosthesis function and the patient's functional abilities after TKA. The KSS clinical evaluation included a questionnaire completed by the investigators to assess for pain, stability, flexion contracture, extension lag, and alignment and evaluated based on number of subjects experiencing any of these issues at the 2-year postoperative visit.
Time Frame: 2 years postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 46 | 46
Participants
  Pain - none | 26 | 27
  Pain - mild or occasional | 12 | 14
  Pain - stairs only | 1 | 1
  Pain - walking & stairs | 1 | 1
  Pain - moderate occasional | 2 | 1
  Pain - moderate continuous | 3 | 1
  Pain - severe | 1 | 0
  Pain - missing response | 0 | 1
  AP Stability - <5 mm | 43 | 43
  AP Stability - 5-10 mm | 1 | 1
  AP Stability - >10 mm | 0 | 1
  AP Stability - missing response | 2 | 1
  Medio-lateral Stability - <6 degrees | 44 | 44
  Medio-lateral Stability - 6-9 degrees | 0 | 0
  Medio-lateral Stability - 10-14 degrees | 0 | 0
  Medio-lateral Stability - >14 degrees | 0 | 1
  Medio-lateral Stability - missing response | 2 | 1
  Flexion Contracture - 0-4 degrees | 42 | 42
  Flexion Contracture - 5-10 degrees | 2 | 2
  Flexion Contracture - 11-15 degrees | 0 | 0
  Flexion Contracture - 16-20 degrees | 0 | 0
  Flexion Contracture - > 20 degrees | 0 | 0
  Flexion Contracture - missing response | 2 | 2
  Extension Lag - 0 degrees | 43 | 44
  Extension Lag - < 10 degrees | 1 | 0
  Extension Lag - 11-20 degrees | 0 | 0
  Extension Lag - > 20 degrees | 0 | 1
  Extension Lag - missing response | 2 | 1
  Alignment - 5 or 10 degrees valgus (normal) | 40 | 41
  Alignment - 4 or 11 degrees valgus | 1 | 1
  Alignment - 3 or 12 degrees valgus | 1 | 1
  Alignment - 2 or 13 degrees valgus | 0 | 0
  Alignment - 1 or 14 degrees valgus | 0 | 1
  Alignment - 0 or 15 degrees valgus | 1 | 0
  Alignment - varus or > 15 degrees valgus | 0 | 0
  Alignment - missing response | 3 | 2

3. Secondary Outcome: Evaluation of Mechanical Alignment Assessed as Either Neutral or Varus/Valgus 3 Months Postoperatively Using a Full Leg X-ray
Description: Long radiographic anterior-posterior (AP) (full-leg standing x-rays) of the entire limb are superior for measuring alignment of the knee as the limb mechanical axes may be more precisely computed. For full-leg x-rays, 2 lines were drawn on the radiograph. First, a line was drawn from the center of the femoral head to the center of the femoral intercondylar notch and the line was extended through to the ankle. Second, a line was drawn from the center of the tibial spine to the center of the ankle talus. The angle between the first and second line was measured to determine mechanical alignment and assessed as either neutral (0 degrees) or a number of degrees of varus or valgus.
Time Frame: 3 months postoperative
Population: Evaluation of Mechanical Alignment 3 Months Postoperatively was not completed for all enrolled subjects. Only data for 88 participants was available.
Measure: Count of Participants; unit: Participants
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 44 | 44
Participants
  Alignment - Neutral | 19 | 10
  Varus | 11 | 28
  Valgus | 14 | 6
  Missing | 0 | 0

4. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Preoperatively and Postoperatively
Description: Evaluation of KOOS questionnaire total scores including categories for symptoms, pain, function of daily living, function of sports and recreational activities, and quality of life. KOOS total scores ranged from 0 to 100, with 0 indicating worst (no function) and 100 indicating no symptoms at all.
Time Frame: Baseline (preoperative), 3 months, 1 year, and 2 years postoperatively
Population: Not all enrolled subjects completed the KOOS questionnaire at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 62 | 60
score on a scale
  Pain - preoperative | 40.9 (17.0) | 43.9 (16.6)
  Pain - 3 months postoperative: number analyzed (Participants) | 58 | 56
  Pain - 3 months postoperative | 73.7 (15.5) | 76.3 (16.1)
  Pain - 1 year postoperative: number analyzed (Participants) | 54 | 49
  Pain - 1 year postoperative | 85.4 (16.7) | 88.5 (16.7)
  Pain - 2 years postoperative: number analyzed (Participants) | 46 | 45
  Pain - 2 years postoperative | 89.4 (13.2) | 92.3 (10.2)
  Symptoms - preoperative: number analyzed (Participants) | 61 | 60
  Symptoms - preoperative | 46.6 (21.2) | 49.9 (17.7)
  Symptoms - 3 months postoperative: number analyzed (Participants) | 58 | 56
  Symptoms - 3 months postoperative | 66.4 (17.5) | 73.1 (13.6)
  Symptoms - 1 year postoperative: number analyzed (Participants) | 54 | 49
  Symptoms - 1 year postoperative | 81.6 (17.2) | 82.5 (16.4)
  Symptoms - 2 years postoperative: number analyzed (Participants) | 45 | 44
  Symptoms - 2 years postoperative | 85.7 (10.9) | 88.2 (9.4)
  Activities of Daily Living (ADLs) - preoperative | 46.5 (18.9) | 51.4 (18.8)
  ADLs - 3 months postoperative: number analyzed (Participants) | 58 | 55
  ADLs - 3 months postoperative | 78.8 (14.6) | 84.1 (13.8)
  ADLs - 1 year postoperative: number analyzed (Participants) | 54 | 49
  ADLs - 1 year postoperative | 86.8 (14.9) | 89.5 (12.4)
  ADLs - 2 years postoperative: number analyzed (Participants) | 46 | 45
  ADLs - 2 years postoperative | 89.3 (14.6) | 92.3 (10.4)
  Sports/Rec - preoperative: number analyzed (Participants) | 58 | 57
  Sports/Rec - preoperative | 19.0 (19.0) | 23.1 (22.8)
  Sports/Rec - 3 months postoperative: number analyzed (Participants) | 44 | 41
  Sports/Rec - 3 months postoperative | 42.4 (29.6) | 48.2 (31.3)
  Sports/Rec - 1 year postoperative: number analyzed (Participants) | 46 | 40
  Sports/Rec - 1 year postoperative | 62.0 (32.0) | 62.5 (32.6)
  Sports/Rec - 2 years postoperative: number analyzed (Participants) | 33 | 36
  Sports/Rec - 2 years postoperative | 74.9 (26.6) | 74.4 (25.6)
  Quality of Life (QoL) - preoperative: number analyzed (Participants) | 62 | 59
  Quality of Life (QoL) - preoperative | 21.0 (17.2) | 22.5 (17.2)
  QoL - 3 months postoperative: number analyzed (Participants) | 58 | 56
  QoL - 3 months postoperative | 58.6 (21.7) | 64.1 (19.9)
  QoL - 1 year postoperative: number analyzed (Participants) | 54 | 49
  QoL - 1 year postoperative | 68.1 (26.2) | 72.9 (23.7)
  QoL - 2 years postoperative: number analyzed (Participants) | 46 | 44
  QoL - 2 years postoperative | 75.1 (23.2) | 78.0 (18.3)

5. Secondary Outcome: Serial Radiographic Evaluations to Assess Evidence of Loosening (Radiolucencies) by Measuring Lucent Zones at 1 Year Postoperatively
Description: X-ray evaluations performed to assess for evidence of implant loosening by radiolucencies (> 2 mm). Anterior-posterior (AP) and lateral serial x-ray evaluations were performed. The span of the bone-prosthesis interface, for each component, was broken down into zone systems. The scoring system for each of the 3 components was determined by measuring the radiolucent lines (mm) for each of these zones.
Time Frame: 1 year postoperatively
Population: Not all subjects completed the serial radiographic evaluations at the specified time points.
Measure: Number; unit: participants
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 54 | 50
participants
  Lucency - femoral zone 1 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 1 (≤ 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 1 (> 2 mm) | 0 | 0
  Lucency - femoral zone 1 (> 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 2 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 2 (≤ 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 2 (> 2 mm) | 0 | 0
  Lucency - femoral zone 2 (> 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 3 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 3 (≤ 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 3 (> 2 mm) | 0 | 0
  Lucency - femoral zone 3 (> 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 4 (≤ 2 mm) | 1 | 0
  Lucency - femoral zone 4 (≤ 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 4 (> 2 mm) | 0 | 0
  Lucency - femoral zone 4 (> 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 5 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 5 (≤ 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 5 (> 2 mm) | 0 | 0
  Lucency - femoral zone 5 (> 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 6 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 6 (≤ 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 6 (> 2 mm) | 0 | 0
  Lucency - femoral zone 6 (> 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 7 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 7 (≤ 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 7 (> 2 mm) | 0 | 0
  Lucency - femoral zone 7 (> 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 1 (≤ 2 mm) | 0 | 0
  Lucency - patellar zone 1 (≤ 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 1 (> 2 mm) | 0 | 0
  Lucency - patellar zone 1 (> 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 2 (≤ 2 mm) | 0 | 0
  Lucency - patellar zone 2 (≤ 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 2 (> 2 mm) | 0 | 0
  Lucency - patellar zone 2 (> 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 3 (≤ 2 mm) | 0 | 0
  Lucency - patellar zone 3 (≤ 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 3 (> 2 mm) | 0 | 0
  Lucency - patellar zone 3 (> 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 4 (≤ 2 mm) | 0 | 0
  Lucency - patellar zone 4 (≤ 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 4 (> 2 mm) | 0 | 0
  Lucency - patellar zone 4 (> 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 5 (≤ 2 mm) | 0 | 0
  Lucency - patellar zone 5 (≤ 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 5 (> 2 mm) | 0 | 0
  Lucency - patellar zone 5 (> 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 6 (≤ 2 mm) | 0 | 0
  Lucency - patellar zone 6 (≤ 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 6 (> 2 mm) | 0 | 0
  Lucency - patellar zone 6 (> 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 7 (≤ 2 mm) | 0 | 0
  Lucency - patellar zone 7 (≤ 2 mm and progressive) | 0 | 0
  Lucency - patellar zone 7 (> 2 mm) | 0 | 0
  Lucency - patellar zone 7 (> 2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 1 (≤ 2 mm) | 3 | 0
  Lucency - tibial AP zone 1 (≤ 2 mm and progressive | 0 | 1
  Lucency - tibial AP zone 1 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 1 (> 2 mm and progressive | 0 | 0
  Lucency - tibial AP zone 2 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 2 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 2 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 2 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 3 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 3 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 3 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 3 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 4 (≤ 2 mm) | 2 | 1
  Lucency - tibial AP zone 4 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 4 (> 2 mm) | 0 | 1
  Lucency - tibial AP zone 4 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 5 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 5 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 5 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 5 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 6 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 6 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 6 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 6 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 7 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 7 (≤2 mm and progressive) | 1 | 0
  Lucency - tibial AP zone 7 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 7 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 8 (≤ 2 mm) | 1 | 0
  Lucency - tibial AP zone 8 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 8 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 8 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 9 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 9 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 9 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 9 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone A (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone A (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone A (> 2 mm) | 0 | 0
  Lucency - tibial AP zone A (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone B (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone B (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone B (> 2 mm) | 0 | 0
  Lucency - tibial AP zone B (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 1 (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone 1 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 1 (> 2 mm) | 0 | 0
  Lucency - tibial ML zone 1 (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 2 (≤ 2 mm) | 1 | 0
  Lucency - tibial ML zone 2 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 2 (> 2 mm) | 0 | 0
  Lucency - tibial ML zone 2 (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 3 (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone 3 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 3 (> 2 mm) | 0 | 0
  Lucency - tibial ML zone 3 (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 4 (≤ 2 mm) | 1 | 0
  Lucency - tibial ML zone 4 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 4 (> 2 mm) | 0 | 0
  Lucency - tibial ML zone 4 (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 5 (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone 5 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 5 (> 2 mm) | 0 | 0
  Lucency - tibial ML zone 5 (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone A (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone A (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone A (> 2 mm) | 0 | 0
  Lucency - tibial ML zone A (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone B (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone B (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone B (> 2 mm) | 0 | 0
  Lucency - tibial ML zone B (>2 mm and progressive) | 0 | 0

6. Secondary Outcome: Radiographic Outcomes to Assess Evidence of Loosening at 1 Year Postoperatively
Description: X-ray evaluations performed to assess for evidence of implant loosening by lack of evidence of surface wear or particulate debris generation, indications of early osteolysis, implant migration, and/or other clinical or radiographic abnormalities. Anterior-posterior (AP) and lateral serial x-ray evaluations were performed.
Time Frame: 1 year postoperatively
Population: Not all subjects completed the serial radiographic evaluations at the specified time points.
Measure: Number; unit: participants
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 54 | 50
participants
  Patella tracking - normal | 53 | 49
  Patella tracking - lateralized | 1 | 0
  Patella tracking - subluxation | 0 | 1
  Patella tracking - dislocation | 0 | 0
  Fixation - Ingrowth | 35 | 32
  Fixation - x-ray unclear | 0 | 1
  Fixation - indifferent, bone unchanged | 34 | 29
  Fixation - increased osseointegration | 1 | 2
  Fixation - bone loss | 0 | 0
  Fixation - implant at risk | 0 | 0
  Fixation - implant loosening | 0 | 0
  Fixation - revision indication | 0 | 0
  Observations - periosteal hypertrophy | 0 | 0
  Observations - osteolysis | 0 | 0
  Observations - subsidence | 0 | 0
  Observations - other | 0 | 0
  Evidence of deformity - no | 54 | 50
  Evidence of deformity - yes | 0 | 0

7. Secondary Outcome: Serial Radiographic Evaluations to Assess Evidence of Loosening at 2 Years Postoperatively
Description: X-ray evaluations performed to assess for evidence of implant loosening by radiolucencies (> 2 mm), lack of evidence of surface wear or particulate debris generation, indications of early osteolysis, implant migration, and/or other clinical or radiographic abnormalities. Anterior-posterior (AP) and lateral serial x-ray evaluations were performed. The span of the bone-prosthesis interface, for each component, was broken down into zone systems. The scoring system for each of the 3 components was determined by measuring the radiolucent lines (mm) for each of these zones.
Time Frame: 2 years postoperatively
Population: Not all subjects completed the serial radiographic evaluations at the specified time points.
Measure: Number; unit: participants
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 45 | 43
participants
  Lucency - femoral zone 1 (≤ 2 mm) | 1 | 0
  Lucency - femoral zone 1 (≤ 2 mm and progressive) | 1 | 0
  Lucency - femoral zone 1 (> 2 mm) | 1 | 0
  Lucency - femoral zone 1 (> 2 mm and progressive) | 0 | 0
  Lucency - femoral zone 2 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 2 (≤2 mm and progressive) | 1 | 0
  Lucency - femoral zone 2 (> 2 mm) | 0 | 0
  Lucency - femoral zone 2 (>2 mm and progressive) | 0 | 0
  Lucency - femoral zone 3 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 3 (≤2 mm and progressive) | 0 | 0
  Lucency - femoral zone 3 (> 2 mm) | 0 | 0
  Lucency - femoral zone 3 (>2 mm and progressive) | 0 | 0
  Lucency - femoral zone 4 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 4 (≤2 mm and progressive) | 0 | 0
  Lucency - femoral zone 4 (> 2 mm) | 0 | 0
  Lucency - femor0al zone 4 (>2 mm and progressive) | 0 | 0
  Lucency - femoral zone 5 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 5 (≤2 mm and progressive) | 0 | 0
  Lucency - femoral zone 5 (> 2 mm) | 0 | 0
  Lucency - femoral zone 5 (>2 mm and progressive) | 0 | 0
  Lucency - femoral zone 6 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 6 (≤2 mm and progressive) | 0 | 0
  Lucency - femoral zone 6 (> 2 mm) | 0 | 0
  Lucency - femoral zone 6 (>2 mm and progressive) | 0 | 0
  Lucency - femoral zone 7 (≤ 2 mm) | 0 | 0
  Lucency - femoral zone 7 (≤2 mm and progressive) | 0 | 0
  Lucency - femoral zone 7 (> 2 mm) | 0 | 0
  Lucency - femoral zone 7 (>2 mm and progressive) | 0 | 0
  Lucency - patella zone 1 (≤ 2 mm) | 0 | 0
  Lucency - patella zone 1 (≤2 mm and progressive) | 0 | 0
  Lucency - patella zone 1 (> 2 mm) | 0 | 0
  Lucency - patella zone 1 (>2 mm and progressive) | 0 | 0
  Lucency - patella zone 2 (≤ 2 mm) | 0 | 0
  Lucency - patella zone 2 (≤2 mm and progressive) | 0 | 0
  Lucency - patella zone 2 (> 2 mm) | 0 | 0
  Lucency - patella zone 2 (>2 mm and progressive) | 0 | 0
  Lucency - patella zone 3 (≤ 2 mm) | 0 | 0
  Lucency - patella zone 3 (≤2 mm and progressive) | 0 | 0
  Lucency - patella zone 3 (> 2 mm) | 0 | 0
  Lucency - patella zone 3 (>2 mm and progressive) | 0 | 0
  Lucency - patella zone 4 (≤ 2 mm) | 0 | 0
  Lucency - patella zone 4 (≤2 mm and progressive) | 0 | 0
  Lucency - patella zone 4 (> 2 mm) | 0 | 0
  Lucency - patella zone 4 (>2 mm and progressive) | 0 | 0
  Lucency - patella zone 5 (≤ 2 mm) | 0 | 0
  Lucency - patella zone 5 (≤2 mm and progressive) | 0 | 0
  Lucency - patella zone 5 (> 2 mm) | 0 | 0
  Lucency - patella zone 5 (>2 mm and progressive) | 0 | 0
  Lucency - patella zone 6 (≤ 2 mm) | 0 | 0
  Lucency - patella zone 6 (≤2 mm and progressive) | 0 | 0
  Lucency - patella zone 6 (> 2 mm) | 0 | 0
  Lucency - patella zone 6 (>2 mm and progressive) | 0 | 0
  Lucency - patella zone 7 (≤ 2 mm) | 0 | 0
  Lucency - patella zone 7 (≤2 mm and progressive) | 0 | 0
  Lucency - patella zone 7 (> 2 mm) | 0 | 0
  Lucency - patella zone 7 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 1 (≤ 2 mm) | 2 | 0
  Lucency - tibial AP zone 1 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 1 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 1 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 2 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 2 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 2 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 2 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 3 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 3 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 3 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 3 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 4 (≤ 2 mm) | 0 | 1
  Lucency - tibial AP zone 4 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 4 (> 2 mm) | 0 | 1
  Lucency - tibial AP zone 4 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 5 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 5 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 5 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 5 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 6 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 6 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 6 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 6 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 7 (≤ 2 mm) | 0 | 1
  Lucency - tibial AP zone 7 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 7 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 7 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 8 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 8 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 8 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 8 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 9 (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone 9 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone 9 (> 2 mm) | 0 | 0
  Lucency - tibial AP zone 9 (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone A (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone A (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone A (> 2 mm) | 0 | 0
  Lucency - tibial AP zone A (>2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone B (≤ 2 mm) | 0 | 0
  Lucency - tibial AP zone B (≤2 mm and progressive) | 0 | 0
  Lucency - tibial AP zone B (> 2 mm) | 0 | 0
  Lucency - tibial AP zone B (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 1 (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone 1 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 1 (> 2 mm) | 0 | 0
  Lucency - tibial ML zone 1 (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 2 (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone 2 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 2 (> 2 mm) | 0 | 0
  Lucency - tibial ML zone 2 (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 3 (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone 3 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 3 (> 2 mm) | 0 | 0
  Lucency - tibial ML zone 3 (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 4 (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone 4 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 4 (> 2 mm) | 0 | 0
  Lucency - tibial ML zone 4 (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 5 (≤ 2 mm) | 0 | 1
  Lucency - tibial ML zone 5 (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone 5 (> 2 mm) | 0 | 0
  Lucency - tibial ML zone 5 (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone A (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone A (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone A (> 2 mm) | 0 | 0
  Lucency - tibial ML zone A (>2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone B (≤ 2 mm) | 0 | 0
  Lucency - tibial ML zone B (≤2 mm and progressive) | 0 | 0
  Lucency - tibial ML zone B (> 2 mm) | 0 | 0
  Lucency - tibial ML zone B (>2 mm and progressive) | 0 | 0

8. Secondary Outcome: Radiographic Outcomes to Assess Evidence of Loosening at 2 Years Postoperatively
Description: as for outcome 6
Time Frame: 2 years postoperatively
Population: Not all subjects completed the serial radiographic evaluations at the specified time points.
Measure: Number; unit: participants
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 45 | 43
participants
  Patella tracking - normal | 42 | 43
  Patella tracking - lateralized | 2 | 0
  Patella tracking - subluxation | 0 | 0
  Patella tracking - dislocation | 0 | 0
  Patella tracking - missing | 1 | 0
  Fixation - fixation/ingrowth | 28 | 24
  Fixation - x-ray unclear | 0 | 0
  Fixation - indifferent, bone unchanged | 27 | 24
  Fixation - increased osseointegration | 0 | 0
  Fixation - bone loss | 0 | 0
  Fixation - implant at risk | 1 | 0
  Fixation - implant loosening | 0 | 0
  Fixation - revision indication | 0 | 0
  Observations - periosteal hypertrophy | 0 | 0
  Observations - osteolysis | 0 | 0
  Observations - subsidence | 0 | 0
  Observations - other | 1 | 0
  Evidence of deformity - no | 45 | 43
  Evidence of deformity - yes | 0 | 0

9. Secondary Outcome: Evaluation of Health Economic Criteria - Surgical Time Details
Description: Analysis of health data captured during and immediately following surgery: anesthesia time, operative time (skin-to-skin), tray setup, duration of operation, blood loss, incision length, number of instrument trays setup, and number of instrument trays used.
Time Frame: During and immediately following surgery
Population: Not all analysis values were available for all enrolled subjects.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 62 | 60
minutes
  Anesthesia time: number analyzed (Participants) | 57 | 54
  Anesthesia time | 128.8 (37.2) | 126.5 (32.8)
  Skin to skin time: number analyzed (Participants) | 57 | 54
  Skin to skin time | 74.9 (23.5) | 75.4 (23.6)
  Tray setup time: number analyzed (Participants) | 61 | 59
  Tray setup time | 16.5 (13.9) | 19.7 (11.7)
  Duration of operation | 110.6 (29.5) | 110.9 (26.8)

10. Secondary Outcome: Evaluation of Health Economic Criteria - Blood Loss
Description: as for outcome 9
Time Frame: During and immediately following surgery
Population: Not all analysis values were available for all enrolled subjects.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 62 | 60
mL | 105.2 (85.1) | 93.8 (39.0)

11. Secondary Outcome: Evaluation of Health Economic Criteria - Incision Length
Description: as for outcome 9
Time Frame: During and immediately following surgery
Population: Not all analysis values were available for all enrolled subjects.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 61 | 59
mm | 153.6 (21.2) | 156.8 (18.4)

12. Secondary Outcome: Evaluation of Health Economic Criteria - Instrument Tray Use
Description: as for outcome 9
Time Frame: During and immediately following surgery
Population: Not all analysis values were available for all enrolled subjects.
Measure: Mean (Standard Deviation); unit: number of trays
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 60 | 59
number of trays
  Instrument trays used in setup | 5.3 (4.2) | 8.2 (2.6)
  Instrument trays used | 5.1 (3.8) | 8.0 (2.6)

13. Secondary Outcome: Evaluation of Health Economic Surgical Criteria
Description: Analysis of health data captured during and immediately following surgery: surgical approach, cut order, final status of posterior cruciate ligament (PCL), and need for perioperative prophylaxis antibiotics.
Time Frame: During and immediately following surgery
Measure: Number; unit: participants
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
Number analyzed (Participants) | 62 | 60
participants
  Surgical approach - medial parapatellar | 58 | 56
  Surgical approach - subvastus | 0 | 0
  Surgical approach - midvastus | 4 | 2
  Surgical approach - lateral parapatellar | 0 | 1
  Surgical approach - other | 0 | 1
  Surgical approach - missing | 0 | 0
  Cut order - distal cut first | 57 | 46
  Cut order - anterior cut first | 5 | 13
  Cut order - tibial cut first | 0 | 1
  Cut order - missing | 0 | 0
  Final status of PCL - excised | 29 | 27
  Final status of PCL - released | 2 | 3
  Final status of PCL - intact | 13 | 15
  Final status of PCL - N/A (PS component used) | 18 | 15
  Final status of PCL - missing | 0 | 0
  Perioperative prophylaxis antibiotics - no | 0 | 0
  Perioperative prophylaxis antibiotics - yes | 62 | 60

ADVERSE EVENTS:
Time Frame: The time of operation through 2 years postoperatively.
Arm/Group | VISIONAIRE Instrumentation | Standard Instrumentation
All-Cause Mortality (participants affected / at risk) | 1/68 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/66
Other Adverse Events (participants affected / at risk) | 43/68 | 38/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VISIONAIRE Instrumentation (N=68) | Standard Instrumentation (N=66)
Chest pain (Cardiac disorders) | 0 (0) | 1 (2)
Confusion (General disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Painful, hot, stiff knee post-op (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stiff knee requiring manipulation under anesthesia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Contralateral TKR (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes (Endocrine disorders) | 1 (1) | 0 (0)
Knee pes tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vascular calcification, right leg popliteal artery (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Decreased ROM left knee secondary to post-op chest infection, unable to do PT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Suspected chest infection 1 week post-op (Infections and infestations) | 0 (0) | 1 (1)
Superficial wound infection (Infections and infestations) | 1 (1) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Post-op wound inflammation, question of stitch reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cancer of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fall on operated knee resulting in pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall - painful knee and wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Right hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Planned left THA (Surgical and medical procedures) | 1 (1) | 0 (0)
Left IT band tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left knee slight clicking sensation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Determined to be not related, resolved.
Wound dehiscence/extruded stitches (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Left knee arthroscopy (Surgical and medical procedures) | 1 (1) | 0 (0)
Bilateral DVT (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Patient fell on buttock, increased left knee discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Right total knee arthroplasty (Surgical and medical procedures) | 1 (1) | 4 (4)
Arterial blood clots due to mitral valve disease; had a TEE (Cardiac disorders) | 0 (0) | 1 (2)
Medial joint line tenderness with certain twisting maneuvers (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical stenosis with cervical DJD (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea postoperatively during hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Left total knee arthroplasty (Surgical and medical procedures) | 1 (1) | 3 (3)
Patient fell and had minor bruising to study knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mild lateral pain by insertion of ITB left study knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bilateral thigh pain, left worse than right (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bilateral trochanteric bursitis - hips (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Left total shoulder replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Painful left knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar laminectomy, fusion of L3-5 and iliac crest bone graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Heart surgery, insertion of mechanical valve in aorta (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgery for bladder prolapse, mesh removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Ascending aortic dissection repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Chest pain, dx stenosis; catheterization and stent placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
L5-S1 lumbar epidural steroid injection (Surgical and medical procedures) | 1 (7) | 0 (0)
Back surgery for back pain (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Removal of prosthesis, left unicompartmental knee arthroplasty revision (Surgical and medical procedures) | 0 (0) | 1 (1)
Bright red blood from rectum and constipation while in hospital (Gastrointestinal disorders) | 1 (1) | 0 (0)
Left knee instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Appendectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Septic knee (Infections and infestations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Re-hospitalization for GI bleed and anemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound dehiscence requiring sutures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthroscopic shoulder debridement and biceps tenolysis (Surgical and medical procedures) | 1 (1) | 0 (0)
Cervical fusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Whipple procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Right carpal tunnel release (Surgical and medical procedures) | 0 (0) | 1 (1)
Moderate effusion requiring aspiration (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Moderate effusion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Effusion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Right distal radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Left distal radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carpal tunnel pain with injection (Nervous system disorders) | 1 (1) | 0 (0)
Right A1 pulley ganglion cyst aspiration (Surgical and medical procedures) | 1 (1) | 0 (0)
Cervical disc decompression and fusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Left knee injection for osteoarthritis (Surgical and medical procedures) | 1 (1) | 0 (0)
Low back/hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DVT secondary to Factor V (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Persistent knee pain after kneeling on study knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mild effusion, aspiration performed (Surgical and medical procedures) | 1 (1) | 0 (0)
Pain and discomfort in left knee due to osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right knee effusion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Left knee effusion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Peroneal and gastrocnemius vein clot at mid-calf (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Repair of left rotator cuff tear (Surgical and medical procedures) | 1 (1) | 0 (0)
Left knee arthroscopy (Surgical and medical procedures) | 0 (0) | 1 (1)
Right knee aspiration due to effusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Right mid-foot pain requiring cortisone injection (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Knee swollen with no erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Patient reported felt feverish post-op (General disorders) | 1 (1) | 0 (0)
Poor ROM (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in left knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sed rate of 27; reference range 0-15 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Skin and tissues around knee seem thick and woody (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Follow up for poor ROM (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fell post-op x2 at home after standing and getting dizzy (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Patellar dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Degenerative arthritis, right knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Atrial fibrillation after elective right TKA (Cardiac disorders) | 1 (3) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Osteoarthritis right shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ischial bursitis on left (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (General disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Follow up for anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swelling post-op right leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Left knee osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Poor ROM right knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Erythema of wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Joint pain left knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right TKA incision tenderness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Knee arthrofibrosis s/p TKA, treated with manipulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Gastritis, with gallballder polys, had cholecystectomy (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonoscopy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cough x2 days (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bilateral leg and foot pain; lumbar degenerative disc disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TKA on contralateral leg (Surgical and medical procedures) | 0 (0) | 1 (1)
Acute blood loss anemia s/p surgery, transfusion not required (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood in stool, suspected hemorrhoid (Gastrointestinal disorders) | 1 (1) | 0 (0)
Left knee w/ mild pain and crepitance (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Degenerative disc disease w/ revision laminectomy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain; dx degenerative disc disease and thoracic sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The major limitation for this study was not reaching the target number of participants needed to achieve target power and statistical analyses leading to uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days